CLINICAL TRIAL: NCT04815538
Title: The Relationship Between Workplace Environment and Metabolic Syndrome in Different Industries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Roshdy Elkhayat, lecturer, Assiut University
Other Study IDs: Metabolic syndrome and work
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Metabolic Syndrome, Protection Against
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- industrial workers: Active workers more than 1 year in petrochemical plant, fertilizer factory , electrical station and food industry
  Interventions: Behavioral: the subscale of Health-Promoting Lifestyle Profile II
- control group: office work unexposed
  Interventions: Behavioral: the subscale of Health-Promoting Lifestyle Profile II

INTERVENTIONS:
Behavioral: the subscale of Health-Promoting Lifestyle Profile II — Nutritional health behavior included the following nine items: "choose a low-fat diet"; "limit the use of sugars"; "eat servings of bread, cereal, and rice"; "eat servings of fruit"; "eat servings of vegetables"; "eat servings of meat, poultry, fish, dietary guidelines
  Other Names: Occupational Physical activity

SUMMARY:
The prevalence of MetS and its components among industrial workers and its risk factors correlates among them and compare them with those in employees from a nonindustrial setting, and explore the influence of different industries on hematological parameters especially WBCs derangement

DETAILED DESCRIPTION:
Metabolic syndrome (MetS), an important risk factor for Cardio Vascular Disease (CVD), is associated with a 2-fold increase in consequences of CVD and 1.5-fold increase in the total mortality . The term MetS refers to a clustering of CVD risk factors including abdominal obesity, high blood pressure, high blood glucose, high levels of blood triglycerides, and low levels of high-density lipoprotein (HDL) cholesterol. An inappropriate lifestyle is one of the most important risk factors for MetS and CVD . Likely, Workplace and working conditions can affect an employee's lifestyle including dietary intake, physical activity, sleep pattern, and their hobbies.

Workplace environment may also affect the occurrence of metabolic syndrome, Air pollution is another risk factor that can increase the risk of metabolic disorders. Recent epidemiological and experimental studies have reported an association between increased level of air pollution with insulin resistance, weight gain, and obesity . Air pollution is higher in some industrial work environments, including those of the gas and petrochemical industries. This may also increase the risk of MetS and CVD among employees of those workplaces. Few studies have assessed the health of employees in industrial workplaces. However, the working conditions of industrial workplace can have a significant impact on the lifestyle and health of employees.

The prevalence of metabolic syndrome has recently been suggested to vary greatly depending on the subject's business category; high prevalence of metabolic syndrome has been reported among the retired, unemployed, bus drivers, university employees, and workers in the agricultural industry , oil industry , and health care sector .

Type of occupation is also important in development of metabolic syndrome. For example, the incidence of metabolic syndrome in the white-collar workers are higher than other male workers. Those with sedentary or shift work carry a higher risk of metabolic syndrome. The incidence of metabolic syndrome is 2.3-fold higher in those working for 10 or more hours per day.

Multiple studies have linked benzene exposure with the abnormality of hematologic parameters, such as the reduction in the counts of white blood cell (WBC), red blood cell (RBC), neutrophil, and lymphocyte, even at low exposure levels (< 1 ppm). A decreased WBC count has been considered as a key clinical sign of benzene-induced hematotoxicity.

However, studies investigating the relationship between work environment and metabolic syndrome in our region are scarce. We therefore, conducted this study to determine the relationship between work environment and metabolic syndrome among a petrochemical workers & non industrial workers.

ELIGIBILITY:
Inclusion Criteria:

* Active workers more than 1 year in selected plants with matched controls from employee of Assiut University.

Exclusion Criteria:

1. Workers who had been working for less than 1 year in their petrochemical plants
2. Workers with self-reported and/or diagnosed carcinomas, hematological diseases, and/or immune diseases.
3. Workers taking any medicine in the preceding 2 weeks affecting lipid profile & blood picture.
4. Workers unwilling to provide biological samples or doing so in insufficient volume.
5. Workers diagnosed MetS and its components before joing the petrochemical industry.
6. Workers with morbid obesity BMI > 40

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: active exposed industrial workers in selected factories
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic Syndrome no. among each group | up to 12 weeks From date of randomization until the date of first documented progression
  MetS was defined according to International Diabetes Federation criteria as: central obesity (defined as waist circumference 90 cm for men and 80 cm for women, plus any two of the following four factors: Raised TG level (150 mg/dl or on treatment for lipid abnormality), reduced HDL cholesterol (¼90 cm for men and >¼80 cm for women and any two of the following four factors: triglycerides >¼150 mg/ dl, reduced HDL cholesterol (<40 mg/dl in men and <50 mg/dl in women or on treatment for lipid abnormality), raised blood pressure (systolic blood pressure 130 mm Hg or diastolic blood pressure 85 mm Hg or on treatment for hypertension),raised fasting plasma glucose (FPG) (FPG100 mg/dl or on treatment for diabetes).
Nutritional health behavior | up to 12 weeks From date of randomization until the date of first documented progression
  nutritional health behavior was obtained using the subscale of Health-Promoting Lifestyle Profile II. Nutritional health behavior included the following nine items: "choose a low-fat diet"; "limit the use of sugars"; "eat servings of bread, cereal, and rice"; "eat servings of fruit"; "eat servings of vegetables"; "eat servings of meat, poultry, fish, dried beans, eggs and nuts"; "eat servings of milk, yogurt or cheese"; "read labels to identify nutrients"; and "eat breakfast." The number of daily servings for each food group was set according to the dietary guidelines, Participants were asked to rate nine items on a four-point Likert scale, ranging from 1 (never) to 4 (routinely). A higher mean score indicated a greater level of participation in nutritional health behavior.

SECONDARY OUTCOMES:
blood sample for Complete blood picture | up to 12 weeks From date of randomization until the date of first documented progression
  5 ml of blood to measure WBCs derangement

REFERENCES:
- [Background] Huang JH, Li RH, Huang SL, Sia HK, Lee SS, Wang WH, Tang FC. Relationships between different types of physical activity and metabolic syndrome among Taiwanese workers. Sci Rep. 2017 Oct 23;7(1):13735. doi: 10.1038/s41598-017-13872-5. PMID 29061986
- [Background] Hidaka T, Hayakawa T, Kakamu T, Kumagai T, Hiruta Y, Hata J, Tsuji M, Fukushima T. Prevalence of Metabolic Syndrome and Its Components among Japanese Workers by Clustered Business Category. PLoS One. 2016 Apr 15;11(4):e0153368. doi: 10.1371/journal.pone.0153368. eCollection 2016. PMID 27082961
- [Background] Jeong HS. The Relationship between Workplace Environment and Metabolic Syndrome. Int J Occup Environ Med. 2018 Oct;9(4):176-183. doi: 10.15171/ijoem.2018.1346. PMID 30325358
- [Background] Clementi EA, Talusan A, Vaidyanathan S, Veerappan A, Mikhail M, Ostrofsky D, Crowley G, Kim JS, Kwon S, Nolan A. Metabolic Syndrome and Air Pollution: A Narrative Review of Their Cardiopulmonary Effects. Toxics. 2019 Jan 30;7(1):6. doi: 10.3390/toxics7010006. PMID 30704059
- [Background] Mini GK, Sarma PS, Thankappan KR. Overweight, the major determinant of metabolic syndrome among industrial workers in Kerala, India: Results of a cross-sectional study. Diabetes Metab Syndr. 2019 Sep-Oct;13(5):3025-3030. doi: 10.1016/j.dsx.2018.07.009. Epub 2018 Jul 17. PMID 30033228
- [Background] Sajid Jabbar A, Ali ET. Impact of Petroleum Exposure on Some Hematological Indices, Interleukin-6, and Inflammatory Markers of Workers at Petroleum Stations in Basra City. J Environ Public Health. 2020 Aug 4;2020:7693891. doi: 10.1155/2020/7693891. eCollection 2020. PMID 32831856